CLINICAL TRIAL: NCT01648491
Title: Autologous Stem Cells for Urinary Incontinence: Single Patient Compassionate Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-204
Record Dates: First submitted 2012-03-08; First posted 2012-07-24 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell treatment (Experimental): Muscle Biopsy and Injection of autologous stem cells
  Interventions: Procedure: Muscle Biopsy; Biological: Injection of autologous stem cells

INTERVENTIONS:
Procedure: Muscle Biopsy — Biopsy of thigh muscle to obtain stem cell core.
Biological: Injection of autologous stem cells — After autologous stem cells have multiplied over 6 weeks time they are injected into the subjects urethra.

SUMMARY:
Determine safety and effectiveness of the technique using autologous stem cells in the treatment of urinary incontinence in one male subject.

DETAILED DESCRIPTION:
Autologous stem cells will be obtained from the subject by needle biopsy, sent to a lab for multiplication and after about 6 weeks time will be injected into the subjects urethra.

ELIGIBILITY:
Inclusion Criteria:

* urinary incontinence
* failed urinary incontinence (UI) treatments

Exclusion Criteria:

- does not meet inclusion criteria, gender and age limit

Ages: 78 Years to 82 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stem Cell Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stem Cell Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Study-Related Adverse Events
Time Frame: 6 months
Measure: Number; unit: Adverse Events
Arm/Group | Stem Cell Treatment
Number analyzed (Participants) | 1
Adverse Events | 0

2. Secondary Outcome: Quality of Life (QOL) Described by the Patient's Response on the Patient Global Assessment of Severity (PGI-S) Questionnaire
Description: The PGI-S is comprised of two questions. Question 1 asks the patient to describe how their urinary tract condition is now. Responses are 1 Normal, 2 Mild, 3 Moderate and 4 Severe. Question 2 asks the patient "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" Responses are 1 Delighted, 2 Pleased, 3 Mostly Satisfied, 4 Mixed, 5 Mostly Dissatisfied, 6 Unhappy and 7 Terrible.
Time Frame: Baseline and 6 months
Measure: Number; unit: units on a scale
Arm/Group | Stem Cell Treatment
Number analyzed (Participants) | 1
units on a scale
  Question 1: Baseline Score | 4
  Question 1: 6 Months Post-Injection Score | 4
  Question 2: Baseline Score | 5
  Question 2: 6 Months Post-Injection Score | 6

3. Secondary Outcome: Quality of Life (QOL) Described by the Patient's Response on the Global Response Assessment (GRA)
Description: The GRA measures overall improvement with therapy. The patient's response describes their current condition compared to before they were treated. Responses are: 1 Markedly Improved, 2 Moderately Improved, 3 Slightly Improved, 4 No Change, 5 Slightly Worse, 6 Moderately Worse, and 7 Markedly Worse.
Time Frame: 6 months
Measure: Number; unit: units on a scale
Groups:
- Stem Cell Treatment: Muscle biopsy and injection of autologous stem cells. Muscle Biopsy: Biopsy of thigh muscle to obtain stem cell core. Injection of autologous stem cells: After autologous stem cells have multiplied over 6 weeks time they are injected into the urethra.
Arm/Group | Stem Cell Treatment
Number analyzed (Participants) | 1
units on a scale | 4

4. Secondary Outcome: Quality of Life (QOL) Described by the Patient's Response on the Patient Global Impression of Improvement (PGI-I)
Description: The PGI-I is a global index used to rate the response of a condition to a therapy. The patient's response describes their current condition compared to before they were treated. Responses are: 1 Very Much Better, 2 Much Better, 3 A Little Better, 4 No Change, 5 A Little Worse, 6 Much Worse, and 7 Very Much Worse.
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | Stem Cell Treatment
Number analyzed (Participants) | 1
units on a scale | 4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Stem Cell Treatment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
This is a single patient compassionate use treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No